CLINICAL TRIAL: NCT01486810
Title: Open-Label Pilot Study of Lisdexamfetamine for Cocaine Dependence
Acronym: Vyvance
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, John Mariani MD, research psychiatrist, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #6154; P50DA009236-18 (NIH)
Record Dates: First submitted 2011-11-30; First posted 2011-12-07 (Estimated); Results first posted 2018-07-11 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Cocaine Dependence
Keywords: cocaine; lisdexamfetamine
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Lisdexamfetamine Dimesylate; Medication Therapy Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lisdexamfetamine and medication management (Experimental): Patients will be titrated to the tolerated dose of Lisdexamfetamine over a two week period, with a maximum of 140mg daily, and then maintained on the highest tolerated dose for four weeks. All participants will receive medication management counseling and individual therapy using a structured compliance enhancement manual designed for pharmacotherapy trials in subjects with substance use disorders.
  Interventions: Drug: Lisdexamfetamine; Behavioral: medication management

INTERVENTIONS:
Drug: Lisdexamfetamine — Patients will be titrated to the tolerated dose over a two week period, with a maximum of 140mg daily, and then maintained on the highest tolerated dose for four weeks
  Other Names: Vyvance
Behavioral: medication management — All participants will receive medication management counseling and individual therapy using a structured compliance enhancement manual designed for pharmacotherapy trials in subjects with substance use disorders.

SUMMARY:
The proposed protocol is an open-label pilot study of the treatment of cocaine dependence using lisdexamfetamine (LDX), a prodrug of d-amphetamine. The investigators plan to enroll 12 patients in an eight-week open-label trial to obtain preliminary data regarding the safety, tolerability, and potential utility of lisdexamfetamine for treatment of cocaine dependence and to determine an effective dosage range.

DETAILED DESCRIPTION:
In an eight-week open label outpatient pilot trial, we will evaluate the safety, tolerability, and potential utility of LDX in the treatment of cocaine dependence. Patients will receive a flexible-fixed dosing schedule under open-label conditions. Patients will be titrated to the tolerated dose over a two week period, with a maximum of 140mg daily, and then maintained on the highest tolerated dose for four weeks, followed by a two week run-down period. All participants will receive medication management counseling and individual therapy using a structured compliance enhancement manual designed for pharmacotherapy trials in subjects with substance use disorders.

The primary outcome measures will be 1) the maximum total lisdexamfetamine dose achieved during the study period defined as the highest amount of medication per day maintained for a seven day period 2) lisdexamfetamine tolerability as measured by adverse effects reported on the Systematic Assessment for Treatment and Emergent Events (SAFTEE). Secondary outcome measures will be 1) cocaine use as recorded by the number of days of use on the Timeline Follow-Back method (Sobell & Sobell, 1992) and confirmed by urine toxicology, 2) cocaine craving as measured by the Cocaine Craving Scale (CCS) and Cocaine Craving Questionnaire (CCQ) and 3) alternate measures of cocaine use, such as the dollar value of cocaine used per day, as measured by the Timeline Follow-Back method, and the proportion of urine toxicology samples negative for cocaine.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must be treatment seeking
* Men and women between the ages of 18-60 who meet DSM-IV criteria for current cocaine dependence
* Used cocaine at least four days in the past month
* Individuals must be in good general health
* Individuals must be capable of giving informed consent and capable of complying with study procedures
* Women of child-bearing age must agree to use a method of contraception with proven efficacy, consisting of one of the following: 1) Any form of hormonal contraception; 2) Intra-uterine device; 3) Sterilization; 4) Double-barrier contraception which is a combination of two of the following: condoms, spermicide, diaphragm. Pregnancy tests will be performed monthly and if a woman becomes pregnant, the study medication will be discontinued.

Exclusion Criteria:

* Individuals who meet DSM-IV-TR criteria for bipolar disorder, schizophrenia, any psychotic disorder other than transient psychosis due to drug abuse, or current major depressive disorder
* Individuals with any other current Axis I psychiatric disorder as defined by DSM-IV-TR that in the investigator's judgment are unstable, or would be disrupted by study medication, or are likely to require pharmacotherapy during the study period
* Individuals physiologically dependent on any other drugs (excluding nicotine or cannabis) which require medical intervention
* Individuals with current psychostimulant abuse or dependence (other than cocaine dependence)
* Individuals with current suicidal risk
* Individuals with coronary vascular disease as indicated by history or suspected by abnormal ECG or history of cardiac symptoms
* Unstable physical disorders which might make participation hazardous such as uncontrolled hypertension (SBP > 140, DBP> 90, or HR > 100 when sitting quietly), acute hepatitis (patients with chronic mildly elevated transaminases < 1.5x upper limit of normal are acceptable), or uncontrolled diabetes
* Individuals with a history of seizures, hyperthyroidism and/or glaucoma
* Individuals with a family history of sudden cardiac death
* History of allergic reaction to study medication
* Women who are pregnant or nursing
* Currently being prescribed psychotropic medication by another physician (other than sleep medication)
* Individuals who are legally mandated (e.g., to avoid incarceration) to participate in substance abuse treatment program

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Mariani, M.D., Principal Investigator — Columbia University
Locations (1):
- STARS, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lisdexamfetamine and Medication Management
Started | 17
Completed | 9
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Lisdexamfetamine and Medication Management
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 3
  More than one race | 3
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Maintained on the Maximum Lisdexamfetamine Daily Dose.
Description: Number of participants achieving and maintained for a seven day period during the trial on the maximum daily dose of 140 mg..
Time Frame: during 1 week of study participation
Population: Although 17 participants were enrolled, one participant was lost to follow-up without any post-enrollment study data, therefore 16 participants were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Lisdexamfetamine and Medication Management
Number analyzed (Participants) | 16
Participants | 12

2. Primary Outcome: Mean Maximum Maintained Dose of Lisdexamfetamine for at Least 1 Week of Trial.
Description: The mean maximum daily dose of lisdexamfetamine that was maintained for at least 1 week of trial.
Time Frame: during 8 weeks of trial or length of participation
Population: data available for 16 participants.
Measure: Mean (Standard Deviation); unit: mgs/day
Arm/Group | Lisdexamfetamine and Medication Management
Number analyzed (Participants) | 16
mgs/day | 118.1 (40.4)

ADVERSE EVENTS:
Arm/Group | Lisdexamfetamine and Medication Management
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 13/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lisdexamfetamine and Medication Management (N=16)
abdominal pain (Gastrointestinal disorders) | 1 (1)
appetite change (General disorders) | 6 (6)
constipation (Gastrointestinal disorders) | 1 (1)
increased heart rate (Cardiac disorders) | 2 (2)
diarrhea (Gastrointestinal disorders) | 2 (2)
dry mouth (General disorders) | 2 (2)
headache (General disorders) | 1 (1)
increased blood pressure (Cardiac disorders) | 1 (1)
insomnia (General disorders) | 3 (3)
jittery (General disorders) | 5 (5)
nausea (Gastrointestinal disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)
fatigue (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
As this was an open label trial, future studies should evaluate lisdexamfetamine for the treatment cocaine use disorder under double-blind conditions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes